CLINICAL TRIAL: NCT06903481
Title: Precision Sleep Medicine: Hardware and Software Innovations for the Combined Diagnosis and Treatment of Sleep Apnea at the Point-of-Care
Brief Title: Precision Sleep Medicine
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Rekonas GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-00175; kt24Herrmann
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Polysomnography (PSG) recordings
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: Adults who underwent polysomnography recordings at the University Hospital Basel in 2023.
- Children and adolescents: Children and adolescents who underwent polysomnography recordings at the University Children's Hospital Basel between January 2022 to July 2024.

SUMMARY:
This retrospective observational study aims to characterize the prevalence and clinical features of obstructive sleep apnea (OSA) phenotypes and develop a rater-independent algorithm for automated OSA phenotyping, improving diagnosis and personalized treatment.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repeated upper airway blockages during sleep, but it presents with a range of phenotypic variations, each with potentially distinct clinical implications. Current clinical definitions are not always precise, making it difficult to clearly classify patients with overlapping features. This phenotypic overlap poses challenges for understanding the true prevalence of "pure" versus "mixed" OSA phenotypes and their respective clinical implications.

To comprehensively characterize the prevalence and clinical features of distinct OSA phenotypes in a large, diverse patient population, this retrospective study analyzes polysomnography (PSG) data from two publicly available National Sleep Research Resource datasets. The findings are then compared to datasets from the University Hospital Basel and University Children's Hospital Basel to assess generalizability.

Furthermore, the study employs computer-aided analysis of PSG data to develop rater-independent algorithms for objective and automated OSA phenotyping. These advancements aim to improve understanding of OSA heterogeneity, facilitating more precise diagnoses and personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* age 19 years and older (data from University Hospital Basel (USB))
* age 18 years or younger (data from University Children's Hospital Basel (UKBB))
* Epworth Sleepiness Scale (ESS) score available (USB only)
* Diagnosis available (e.g. Obstructive sleep apnea (OSA), Central Sleep Apnea (CSA), Cheyne Stokes Breathing (CSR), ...)
* signed written general consent

Exclusion Criteria:

* history of treatment of sleep apnea
* tracheostomy
* current home oxygen therapy
* decline to sign the written general consent, or absence of written general consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults who underwent polysomnography recordings at the University Hospital Basel in 2023, as well as children and adolescents who underwent polysomnography recordings at the University Children's Hospital Basel between January 2022 and July 2024. All patients have signed the general consent of the university hospital (UBS), resp. The university children's hospital (UKBB).
Sampling Method: Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Phenotype characterization | 2025
  To characterize the prevalence and clinical features of distinct obstructive sleep apnea (OSA) phenotypes in a large, diverse patient population, polysomnography (PSG) recordings from two publicly available National Sleep Research Resource data collections are analyzed and compared to datasets from the University Hospital Basel (USB) and University Children's Hospital Basel (UKBB) to assess generalizability.

SECONDARY OUTCOMES:
Computer-aided phenotyping | 2025
  To evaluate the potential of computer-aided pattern recognition in improving the accuracy and efficiency of OSA phenotype identification from PSG data, an algorithm is developed that objectively and automatically identifies OSA phenotypes from PSG recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Herrmann, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - University Children's Hospital Basel, Basel, Canton of Basel-City
  - University Hospital Basel, Basel, Canton of Basel-City